CLINICAL TRIAL: NCT05416242
Title: Evaluation of Patient-centered Outcomes Associated With Acceleration of Lower Incisors Decrowding Using Self-ligating Brackets With and Without Piezocision in Comparison With Traditional Brackets: A Randomized Controlled Clinical Trial
Brief Title: Patient-centered Outcomes During Using Self-ligating Brackets With or Without Piezocision vs Traditional Brackets
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Ortho-11-2022
Record Dates: First submitted 2022-06-05; First posted 2022-06-13 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Crowding, Tooth
Keywords: Self-Ligating Brackets; Flapless corticotomy; Severe crowding; Leveling; Aligning
MeSH Terms: conditions — Malocclusion; Crowding

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fixed appliance (Active Comparator): Patients in this group will be treated using traditional brackets alone.
  Interventions: Device: Traditional braces
- Self-ligaton appliance (Experimental): Patients in this group will be treated using self-ligating brackets alone.
  Interventions: Device: Self-ligating braces
- Self-ligaton appliance + piezocision (Experimental): Patients in this group will be treated using self-ligating brackets associated with piezocision.
  Interventions: Procedure: Self-ligating braces + piezocision

INTERVENTIONS:
Device: Traditional braces — MBT 0.022 perception traditional braces will be used without any acceleration method.
  Arms: Fixed appliance
Device: Self-ligating braces — MBT 0.022 perception Self-ligating braces will be used without any acceleration method.
  Arms: Self-ligaton appliance
Procedure: Self-ligating braces + piezocision — Flapless corticotomy will be applied for the upper anterior teeth.
  Arms: Self-ligaton appliance + piezocision

SUMMARY:
The different types of brackets (e.g., self-ligating and conventional brackets), and the various acceleration methods (e.g., corticotomy) cause varying degrees of pain and discomfort. This study will assess pain, discomfort, and other patient-centered outcomes in adults with severe crowding on the upper jaw requiring two first premolars extraction.

There are three groups:

The first group (control group): the patients in this group will be treated using conventional brackets alone.

The second group (Experimental group): the patients in this group will be treated using self-ligating brackets alone.

The third group (Experimental group): the patients in this group will be treated using self-ligating brackets associated with flapless corticotomy.

DETAILED DESCRIPTION:
Pain associated with orthodontic treatment is one of the undesirable complications, which negatively affects the patient's cooperation. Pain may occur due to the pressure on the periodontal ligaments induced by orthodontic forces. The perception of pain is affected by many factors related to the patient, such as age, gender and any previous treatment experiences, which are negatively or positively reflected on the patient's cooperation. As for the factors related to the type of orthodontic treatment provided, the pain and discomfort are proportional to the brackets system used and the forces applied, especially in the leveling and alignment stage. The amount of tooth movement is directly affected by the friction between the brackets and the wires used. The physical properties of the wire and brackets used and the dimensions of the applied wires, in addition to the type of ligation play a significant role in the amount of friction generated.

ELIGIBILITY:
Inclusion Criteria:

1. The patient's age is between 18 and 25 years
2. Severe crowding on the upper jaw (more than 6 mm) requires upper first premolars extraction
3. Little's Index of Irregularity is greater than 7 mm
4. Overbite ranging between 0-4 mm
5. Normal inclination of the upper incisors
6. No missing teeth (except for third molars)
7. Class I or class II (ANB ≤ 5) or class III (ANB ≥ 0)

Exclusion Criteria:

1. The presence of any systemic disease affecting orthodontic movement
2. The presence of congenital syndromes or cleft lip and palate
3. Poor oral health with a plaque index greater than (1)
4. Skeletal maxillary constriction

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2019-04-14 (Actual); Primary Completion 2020-10-07 (Actual); Study Completion 2021-08-22 (Actual)

PRIMARY OUTCOMES:
Change in the levels of pain | After 24 hours; 4 days; 7 days; 14 days; 28 days
  Patients will be asked this question about their feeling of pain (Item no 01):
  'What is the degree of pain you have experienced?' A standardized questionnaire will be used to assess pain, discomfort and functional impairments' levels during the active phase of treatment. The patient will be asked to specify a point on the visual analogue scale (VAS), a 100-mm horizontal line with two focal points at its beginning and end (0: there is no pain - 100: the worst pain). The score will be determined by measuring the distance from the beginning until the point identified by the patient.
Change in the levels of discomfort | After 24 hours; 4 days; 7 days; 14 days; 28 days
  Patients will be asked this question about their feeling of discomfort (Item no 02):
  'What is the degree of discomfort you have experienced?' A standardized questionnaire will be used to assess pain, discomfort and functional impairments' levels during the active phase of treatment. The patient will be asked to specify a point on the visual analogue scale (VAS), a 100-mm horizontal line with two focal points at its beginning and end (0: there is no pain - 100: the worst pain). The score will be determined by measuring the distance from the beginning until the point identified by the patient.
Change in the Perception of swelling | After 24 hours; 4 days; 7 days; 14 days; 28 days
  Patients will be asked this question about their feeling of swelling (Item no 03):
  'What is the degree of swelling you have experienced?' A standardized questionnaire will be used to assess pain, discomfort and functional impairments' levels during the active phase of treatment. The patient will be asked to specify a point on the visual analogue scale (VAS), a 100-mm horizontal line with two focal points at its beginning and end (0: there is no pain - 100: the worst pain). The score will be determined by measuring the distance from the beginning until the point identified by the patient.
Change in the difficulty of mastication | After 24 hours; 4 days; 7 days; 14 days; 28 days
  'What is the degree of mastication difficulties you have experienced?' A standardized questionnaire will be used to assess pain, discomfort and functional impairments' levels during the active phase of treatment. The patient will be asked to specify a point on the visual analogue scale (VAS), a 100-mm horizontal line with two focal points at its beginning and end (0: there is no pain - 100: the worst pain). The score will be determined by measuring the distance from the beginning until the point identified by the patient.
Change in the difficulty of swallowing | After 24 hours; 4 days; 7 days; 14 days; 28 days
  Patients will be asked this question about their feeling of swallowing (Item no 05):
  'What is the degree of swallowing difficulties you have experienced?' A standardized questionnaire will be used to assess pain, discomfort and functional impairments' levels during the active phase of treatment. The patient will be asked to specify a point on the visual analogue scale (VAS), a 100-mm horizontal line with two focal points at its beginning and end (0: there is no pain - 100: the worst pain). The score will be determined by measuring the distance from the beginning until the point identified by the patient.
Change in the perception of the jaw movement restriction | After 24 hours; 4 days; 7 days; 14 days; 28 days
  Patients will be asked this question about their feeling of the jaw movement restriction (Item no 06):
  'What is the degree of the jaw movement restriction you have experienced?' A standardized questionnaire will be used to assess pain, discomfort and functional impairments' levels during the active phase of treatment. The patient will be asked to specify a point on the visual analogue scale (VAS), a 100-mm horizontal line with two focal points at its beginning and end (0: there is no pain - 100: the worst pain). The score will be determined by measuring the distance from the beginning until the point identified by the patient.
The levels of satisfaction | This outcome will be assessed at 28 days following the beginning of treatment
  Patients will be asked this question about their levels of satisfaction (Item no 07): 'What is your levels of satisfaction on the orthodontic treatment provided?' A standardized questionnaire will be used to assess pain, discomfort and functional impairments' levels during the active phase of treatment. The patient will be asked to specify a point on the visual analogue scale (VAS), a 100-mm horizontal line with two focal points at its beginning and end (0: there is no satisfaction- 100: the highest satisfaction). The score will be determined by measuring the distance from the beginning until the point identified by the patient.
Recommendation of the procedure to a friend | This outcome will be assessed at 28 days following the beginning of treatment
  Patients will be asked this question (Item no 08): 'Would you recommend a friend undergo this treatment?' Assessment will be performed using a two-point scale to answer yes or no.
The possibility of repeating the procedure | This outcome will be assessed at 28 days following the beginning of treatment
  Patients will be asked this question about the possibility of repeating the procedure (Item no 09): 'Would you accept to undergo this treatment again?' Assessment will be performed using a two-point scale to answer yes or no.

CONTACTS AND LOCATIONS:
Overall Officials: Heba M Al-Ibrahim, DDS,MSc, Principal Investigator — Department of orthodontics, Damascus University, Syria; Mohammad Y Hajeer, DDS,MSc,PhD, Study Director — Professor of Orthodontics, University of Damascus Dental School, Damascus, Syria.; Issam ِAlkhoury, DDS,MSc,PhD, Study Director — Professor of Oral and Maxillofacial Surgery, University of Damascus Dental School, Damascus, Syria
Locations (1):
- University of Damascus, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jahanbin A, Hasanzadeh N, Khaki S, Shafaee H. Comparison of self-ligating Damon3 and conventional MBT brackets regarding alignment efficiency and pain experience: A randomized clinical trial. J Dent Res Dent Clin Dent Prospects. 2019 Fall;13(4):281-288. doi: 10.15171/joddd.2019.043. PMID 32190212
- [Background] Fleming PS, Dibiase AT, Sarri G, Lee RT. Pain experience during initial alignment with a self-ligating and a conventional fixed orthodontic appliance system. A randomized controlled clinical trial. Angle Orthod. 2009 Jan;79(1):46-50. doi: 10.2319/121007-579.1. PMID 19123718
- [Background] Gibreal O, Hajeer MY, Brad B. Evaluation of the levels of pain and discomfort of piezocision-assisted flapless corticotomy when treating severely crowded lower anterior teeth: a single-center, randomized controlled clinical trial. BMC Oral Health. 2019 Apr 16;19(1):57. doi: 10.1186/s12903-019-0758-9. PMID 30991984
- [Background] Lai TT, Chiou JY, Lai TC, Chen T, Wang HY, Li CH, Chen MH. Perceived pain for orthodontic patients with conventional brackets or self-ligating brackets over 1 month period: A single-center, randomized controlled clinical trial. J Formos Med Assoc. 2020 Jan;119(1 Pt 2):282-289. doi: 10.1016/j.jfma.2019.05.014. Epub 2019 Jun 14. PMID 31208826
- [Background] Tecco S, D'Attilio M, Tete S, Festa F. Prevalence and type of pain during conventional and self-ligating orthodontic treatment. Eur J Orthod. 2009 Aug;31(4):380-4. doi: 10.1093/ejo/cjp003. Epub 2009 May 22. PMID 19465738